CLINICAL TRIAL: NCT03540641
Title: Effect of the Transcranial Magnetic Stimulation Applied on the Left Dorsolateral Prefrontal Cortex on the Clinical and Neuropsychological Variables in Subjects With Binge Eating Disorder
Brief Title: Transcranial Magnetic Stimulation (TMS) in Binge Eating Disorder (BED)
Acronym: TMS&BED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Queretaro (Other)
Responsible Party: Principal Investigator, Dr. Julian Reyes López, professor, Universidad Autonoma de Queretaro
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 9320
Record Dates: First submitted 2018-04-30; First posted 2018-05-30 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Binge-Eating Disorder
Keywords: Binge Eating Disorder; Transcranial Magnetic Stimulation; Food Craving
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1500 pulses (Active Comparator): This group will receive 1500 pulses of transcranial magnetic stimulation at 5Hz over the left dorsolateral prefrontal cortex, until completing 15 sessions
  Interventions: Device: MagVenture MagPro R30
- 1500 pulses sham (Sham Comparator): this group will receive the sham modality of the protocol of 1500 pulses at 5Hz of transcranial magnetic stimulation during 15 sessions.
  Interventions: Device: MagVenture MagPro R30
- 5000 pulses (Active Comparator): This group will receive 5000 pulses of transcranial magnetic stimulation at 5Hz over the left dorsolateral prefrontal cortex, until completing 15 sessions.
  Interventions: Device: MagVenture MagPro R30
- 5000 pulses sham (Sham Comparator): this group will receive the sham modality of the protocol of 5000 pulses at 5Hz of transcranial magnetic stimulation during 15 sessions.
  Interventions: Device: MagVenture MagPro R30

INTERVENTIONS:
Device: MagVenture MagPro R30 — the subjects will receive 1500 or 5000 pulses at 5Hz
  Other Names: repetitive Transcranial Magnetic Stimulation

SUMMARY:
This study evaluates de efficacy of 5Hz repetitive Transcranial Magnetic Stimulation (rTMS) applied on the left dorsolateral prefrontal cortex in patients with binge eating disorder.

DETAILED DESCRIPTION:
Binge Eating Disorder (BED) affects a significant percentage of de national population (1.4%) in a portio 2-1 in woman compared with men, the repetitive Transcranial Magnetic Stimulation (rTMS) is a neuromodulation technique, which allows us to induce brain electrical activity by plating magnetic fields and it has been proven that at 10Hz it has an effect of improvement in the craving of food.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of both sexes.
2. Subjects from 18 to 45 years of age.
3. Subjects with diagnosis of binge eating disorder.
4. Subjects without changes in pharmacological treatment in the last 30 days.
5. Subjects who agree to sign the informed consent letter.

Exclusion Criteria:

1.Subjects with a history of traumatic brain injury with loss of consciousness. 2.Subjects with intracranial metallic objects or metal plates in the skull.

3.Subjects who suffer chronic diseases not controlled at the time of entering the study (for example: hypertension, diabetes, rheumatic diseases).

4.Patients with psychotic symptoms, bipolar affective disorders and substance dependence.

5.Subjects with alterations in electroencephalogram (epileptiform activity). 6.Patients with any type of chronic or neurological medical disease not controlled.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Food Craving Inventory (FCI) | 6 weeks
  The FCI is a self-report inventory designed to measure the food craving, is made up of 37 elements and is a scale-likert instrument.

SECONDARY OUTCOMES:
Barratt Impulsivity Scale (BIS-11) | 6 weeks
  The Barratt Impulsiveness Scale is a questionnaire designed to assess the personality / behavioral construct of impulsiveness is composed of 30 items describing common impulsive or non-impulsive (for reversed scored items) behaviors and preferences .

CONTACTS AND LOCATIONS:
Overall Officials: Julian Reyes López, Doctor, Study Director — Universidad Autónoma de Querétaro
Locations (1):
- Sofía Cañizares Gómez., Querétaro City, Querétaro, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Amianto F, Ottone L, Abbate Daga G, Fassino S. Binge-eating disorder diagnosis and treatment: a recap in front of DSM-5. BMC Psychiatry. 2015 Apr 3;15:70. doi: 10.1186/s12888-015-0445-6. PMID 25885566
- [Result] Orozco-Cabal LF, Herin D. Neurobiologia de la impulsividad y los trastornos de la conducta alimentaria. Rev Colomb Psiquiatr. 2008 Jun 1;37(2):207-219. Spanish. PMID 19838321
- [Result] Maranhao MF, Estella NM, Cury ME, Amigo VL, Picasso CM, Berberian A, Campbell I, Schmidt U, Claudino AM. The effects of repetitive transcranial magnetic stimulation in obese females with binge eating disorder: a protocol for a double-blinded, randomized, sham-controlled trial. BMC Psychiatry. 2015 Aug 12;15:194. doi: 10.1186/s12888-015-0569-8. PMID 26265452
- [Result] Van den Eynde F, Claudino AM, Mogg A, Horrell L, Stahl D, Ribeiro W, Uher R, Campbell I, Schmidt U. Repetitive transcranial magnetic stimulation reduces cue-induced food craving in bulimic disorders. Biol Psychiatry. 2010 Apr 15;67(8):793-5. doi: 10.1016/j.biopsych.2009.11.023. Epub 2010 Jan 8. PMID 20060105
- [Result] Uher R, Rutter M. Classification of feeding and eating disorders: review of evidence and proposals for ICD-11. World Psychiatry. 2012 Jun;11(2):80-92. doi: 10.1016/j.wpsyc.2012.05.005. PMID 22654933
- [Result] Barth KS, Rydin-Gray S, Kose S, Borckardt JJ, O'Neil PM, Shaw D, Madan A, Budak A, George MS. Food cravings and the effects of left prefrontal repetitive transcranial magnetic stimulation using an improved sham condition. Front Psychiatry. 2011 Mar 14;2:9. doi: 10.3389/fpsyt.2011.00009. eCollection 2011. PMID 21556279
- [Result] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472